CLINICAL TRIAL: NCT03886831
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation, Dose Expansion Study of PRT543 in Patients With Advanced Solid Tumors and Hematologic Malignancies
Brief Title: A Study of PRT543 in Participants With Advanced Solid Tumors and Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT543-01
Record Dates: First submitted 2019-03-08; First posted 2019-03-22 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Relapsed/Refractory Advanced Solid Tumors; Relapsed/Refractory Diffuse Large B-cell Lymphoma; Relapsed/Refractory Myelodysplasia; Relapsed/Refractory Myelofibrosis; Adenoid Cystic Carcinoma; Relapsed/Refractory Mantle Cell Lymphoma; Relapsed/Refractory Acute Myeloid Leukemia; Refractory Chronic Myelomonocytic Leukemia
Keywords: PRMT5; PRMT5 Inhibitor
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse; Anemia, Refractory, with Excess of Blasts; Primary Myelofibrosis; Carcinoma, Adenoid Cystic; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT543 (Experimental): PRT543 will be administered orally
  Interventions: Drug: PRT543

INTERVENTIONS:
Drug: PRT543 — PRT543 will be administered orally

SUMMARY:
This is a Phase 1 cohort, dose-escalation, dose-expansion study of PRT543 in patients with advanced cancers who have exhausted available treatment options. The purpose of this study is to define a safe dose and schedule to be used in subsequent development of PRT543.

DETAILED DESCRIPTION:
This is a multicenter, open-label, sequential-cohort, dose-escalation, dose-expansion Phase 1 study of PRT543 in patients with advanced cancers who have exhausted available treatment options. Enrollment will take place concurrently into two distinct patient groups (one for solid tumors/lymphomas and one for hematological malignancies). The study will consist of 2 parts, a dose escalation part, and once the recommended phase 2 dose (RP2D) has been determined, a cohort expansion part involving up to ten separate cohorts. For patients, the study will include a screening phase, a treatment phase, and a post treatment follow-up phase. An end-of-study visit will be conducted within 30 days after the last dose of PRT543.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or advanced solid tumor; or advanced diffuse large B-cell lymphoma; or advanced mantle cell lymphoma; or relapsed myelodysplastic syndrome, acute myeloid leukemia or chronic myelomonocytic leukemia; or relapsed myelofibrosis. All malignancies must be refractory to established therapies
* Biomarker-selected solid tumors
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
* Adequate organ function (bone marrow, hepatic, renal, cardiovascular)
* Female patients of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment and must agree to use an effective method of contraception during the trial

Exclusion Criteria:

* Primary malignancies of the Central Nervous System(CNS) or uncontrolled CNS metastases
* Requirement of pharmacologic doses of glucocorticoids
* Prior treatment with chimeric antigen receptor T cells (CAR-T cells)
* HIV positive; known active hepatitis B or C
* Known hypersensitivity to any of the components of PRT543
* Prior allogeneic bone marrow transplant; autologous hematopoietic transplantation less than 100 days since transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
To describe dose limiting toxicities (DLT) of PRT543 | Baseline through Day 28.
  Dose limiting toxicities (DLTs) will be evaluated during the first cycle
To determine the maximally tolerated dose (MTD) | Baseline through approximately 2 years.
  The maximum tolerated dose (MTD) will be established for further investigation in participants with advanced malignancies who have failed prior treatments.
To determine the recommended phase 2 dose (RP2D) and schedule of PRT543 | Baseline through approximately 2 years.
  The recommended phase 2 dose (RP2D) and optimal dosing schedule of PRT543 will be established for further investigation in participants with advanced malignancies who have failed prior treatments.

SECONDARY OUTCOMES:
To describe the adverse event profile and tolerability of PRT543 | Baseline through approximately 2 years
  Adverse events as characterized by type, frequency, severity, timing, seriousness and relationship to study therapy
To determine the maximum observed plasma concentration (Cmax) of PRT543 | Cycle 1 (each cycle is 28 days) on Days 1, 15, and/or 25: predose and 0.5, 1, 2, 4, 8, 24 hours postdose; predose on Cycle 1, Days 3, 4, 8, 11, and/or 22. Subsequently for Cycle 2 and beyond (until end of study treatment) on Day 1.
  PRT543 pharmacokinetics will be calculated including the maximum observed plasma concentration.
To determine the time to reach maximum observed plasma concentration (Tmax) of PRT543 | Cycle 1 (each cycle is 28 days) on Days 1, 15, and/or 25: predose and 0.5, 1, 2, 4, 8, 24 hours postdose; predose on Cycle 1, Days 3, 4, 8, 11, and/or 22. Subsequently for Cycle 2 and beyond (until end of study treatment) on Day 1.
  PRT543 pharmacokinetics will be calculated including the time to reach maximum observed plasma concentration

OTHER OUTCOMES:
To determine the terminal elimination half-life (t1/2) of PRT543. | Cycle 1 (each cycle is 28 days) on Days 1, 15, and/or 25: predose on Cycle 1, Days 3, 4, 8, 11, and/or 22. Subsequently for Cycle 2 and beyond (until end of study treatment) on Day 1.
  PRT543 pharmacokinetics will be calculated including the terminal elimination half life
To determine the area under the plasma concentration versus time curve (AUC) of PRT543 | Cycle 1 (each cycle is 28 days) on Days 1, 15, and/or 25: predose on Cycle 1, Days 3, 4, 8, 11, and/or 22. Subsequently for Cycle 2 and beyond (until end of study treatment) on Day 1.
  PRT543 pharmacokinetics will be calculated including area under the plasma concentration versus time curve.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UCSF Precision Cancer Medicine Building, San Francisco, California
  - Christiana Care Health Services, Christiana Hospital, Newark, Delaware
  - Florida Cancer Specialists, Lake Mary, Florida
  - Florida Cancer Specialist, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University and Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington